CLINICAL TRIAL: NCT05088174
Title: A Single-Center, Single-Arm, Open-Label, Self-Controlled, Drug-Drug Interaction Study of Hetrombopag Olamine and Ciclosporin in Healthy Subjects
Brief Title: A Trial of Hetrombopag in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR8735-111
Record Dates: First submitted 2021-10-12; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Sever Aplastic Anaemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D1：hetrombopag single dose，D11-D15：cyclosporine,D16 combination use of hetrombopag and cyclosporine (Experimental)
  Interventions: Drug: Hetrombopag Olamine Tablet；Ciclosporin Soft Capsule

INTERVENTIONS:
Drug: Hetrombopag Olamine Tablet；Ciclosporin Soft Capsule — Drug:
  Hetrombopag Olamine Tablet Ciclosporin Soft Capsule

SUMMARY:
This is a single-center, single-arm, open-label, self-controlled, phase I clinical study. A total of 26 male or female healthy subjects are intended to be enrolled to evaluate the PK drug-drug interaction between ciclosporin and hetrombopag.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form prior to any study-related activities, understand the procedures and methods of the study, and agree to complete this study in strict accordance with the clinical study protocol;
2. Male or female subjects aged 18-55 years (inclusive);
3. Body mass index (BMI) between 18 and 26 kg/m2 (inclusive);
4. Normal or abnormal but not clinically significant physical examination and laboratory test results; normal or abnormal but not clinically significant ECG;
5. Have no plan for pregnancy and agree to take effective contraceptive measures from signing of informed consent form until 6 months after the last dose;
6. Able to maintain a consistency of good communication with the investigators, and understand and comply with all the requirements of this study

Exclusion Criteria:

1. Any previous or current serious clinical conditions of the circulatory system, endocrine system, nervous system, digestive system, respiratory system, and hematological, immunological, psychiatric and metabolic abnormalities, or any disease that may interfere with the results of this study;
2. History of deep venous thrombosis or other thrombotic disorders;
3. QTc > 450 ms in males or QTc > 460 ms in females through 12-lead ECG examination with clinical significance per the investigator's judgment at screening;
4. Positive for hepatitis B surface antigen, hepatitis C antibody, syphilis antibody (trust), or HIV antibody;
5. Positive pregnancy test result;
6. Allergic constitution, or allergy to any component of hetrombopag olamine tablets and ciclosporin capsules;
7. Have received surgery within 4 weeks before the first study administration, or plan to undergo surgery during the course of the study;
8. Have taken any drug that alters liver enzyme activity within 28 days before the first study administration or during the study;
9. Have taken any prescription drug, over-the-counter drug, herbal medicine, or health supplements within 14 days before the first study administration, or within 5 half-lives of the drug at screening; plan to take non-study drugs or health supplements during the study;
10. Consumption of grapefruit or grapefruit-containing products, foods or beverages containing caffeine, xanthine, or alcohol within 48 h before the first study administration; strenuous exercise, or other factors that affect drug absorption, distribution, metabolism, and excretion;
11. Have participated in any drug clinical trial and have been treated with any investigational drug or medical device within 3 months before the first study administration (per the date of signing the informed consent form);
12. Have blood donation (or blood loss) of ≥ 400 mL or have received blood transfusion within 3 months before screening;
13. Unable or unwilling to comply with the lifestyle requirements in the protocol;
14. Addicted to smoking (≥ 5 cigarettes per day within 1 month before screening);
15. Average daily alcohol consumption of > 15 g for females (e.g., 145 mL of wine, 497 mL of beer, or 43 mL of low-alcohol liquor) and > 25 g for males (e.g., 290 mL of wine, 994 mL of beer, or 86 mL of low-alcohol liquor) within 1 month before screening;
16. History of drug abuse, history of drug dependence, or drug abuse screening positive (drugs include morphine, methamphetamine, ketamine, ecstasy (dimethylene dioxyamphetamine), and cannabis (tetrahydrocannabinol)) (consultation and examination), or history of drug abuse within the past five years or have used narcotics within 3 months before the study;
17. Potentially unable to complete the study for other reasons or judged by the investigator as not suitable for the study.
18. Intolerant to venipuncture, or history of hemophobia or fear of needles;
19. Have special dietary requirements and unable to accept a standardized diet;
20. Acute disease from screening to first study administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Peak hetrombopag plasma concentration (Cmax) | 0-120 hours post dose
Area Under the plasma hetrombopag concentration vs time curve (AUC0-120) | 0-120 hours post dose
Area under the plasma hetrombopag concentration vs time curve (AUC0-inf) | 0-infinity

SECONDARY OUTCOMES:
Time to Reach Maximum Drug Concentration in Plasma After Single Dose (Tmax) | 0-120 hours post dose
Half-life Associated With the Terminal Slope (t½) | 0-120 hours post dose
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 22

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital Ethics Committee, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided